CLINICAL TRIAL: NCT00017316
Title: A Phase II, Pharmacologic and Biologic Study of Escalating Doses of Thalidomide (NSC #66847) Administered Orally Once a Day in Combination With a Fixed Dose of SU5416 (NSC #696819) in Patients With Metastatic Melanoma
Brief Title: Thalidomide and SU5416 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068677; UTHSC-IDD-99-27; SACI-IDD-99-27; NCI-66
Record Dates: First submitted 2001-06-06; First posted 2003-06-12 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2002-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Semaxinib; Thalidomide

ARMS (1):
- Arm I (Experimental): Patients receive SU5416 IV over 1 hour twice weekly and oral thalidomide daily beginning 1 day after the first dose of SU5416. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: semaxanib; Drug: thalidomide

INTERVENTIONS:
Drug: semaxanib
Drug: thalidomide

SUMMARY:
Phase II trial to study the effectiveness of combining thalidomide and SU5416 in treating patients who have metastatic melanoma. Thalidomide combined with SU5416 may stop the growth of metastatic melanoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of thalidomide and SU5416 in patients with metastatic melanoma.

II. Determine the quantitative and qualitative toxic effects of this regimen in these patients.

III. Evaluate the pharmacokinetics of this regimen in these patients. IV. Determine the complete and partial responses and response duration in patients treated with this regimen.

V. Assess disease-free survival at 6 months of patients treated with this regimen.

OUTLINE:

Patients receive SU5416 IV over 1 hour twice weekly and oral thalidomide daily beginning 1 day after the first dose of SU5416. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic melanoma
* Bidimensionally measurable disease by MRI, CT scan, or chest x-ray
* No active brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.5 g/dL

Hepatic:

* PT/PTT normal
* Bilirubin no greater than 1.5 mg/dL
* SGOT/SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No uncompensated coronary artery disease by electrocardiogram or physical exam
* No myocardial infarction or severe or unstable angina within the past 6 months
* No deep venous thrombosis within the past 3 months
* No arterial thrombosis within the past 6 months

Pulmonary:

* No pulmonary embolism within the past 6 months

Other:

* HIV negative
* No active infection
* No medical, psychological, or social problem that would preclude study participation
* No history of gastrointestinal disorder that would interfere with absorption or swallowing of study medication
* No emotional disorder or substance abuse
* No diabetes mellitus with severe peripheral vascular disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 4 weeks before, during, and for 4 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior biologic regimen
* No concurrent biologic response modifiers
* No concurrent hematopoietic growth factor support
* Concurrent epoetin alfa allowed

Chemotherapy:

* No concurrent cytotoxic agents

Endocrine therapy:

* No concurrent anticancer hormonal therapy except megestrol acetate for appetite stimulation

Radiotherapy:

* No prior large field radiotherapy to more than 20% total bone marrow
* No concurrent radiotherapy

Surgery:

* At least 14 days since major surgery
* No prior major upper gastrointestinal surgery

Other:

* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-03; Primary Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States